CLINICAL TRIAL: NCT04002414
Title: Physical Activity and Fertility Care Study
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-28431
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Infertility, Female
Keywords: Physical Activity; In Vitro Fertilization; Ovarian Stimulation; Exercise
MeSH Terms: conditions — Infertility, Female; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be stratified into groups: "active" or "insufficiently active" based on current average physical activity. Randomization will be into one of two parallel arms, maintenance of current activity during ovarian stimulation, or modify activity level during ovarian stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usually Active- Decrease (Active Comparator): Participants who usually meet or exceed recommended levels of physical activity who will be asked to minimize activity during stimulation.
  Interventions: Behavioral: Insufficient physical activity
- Usually Active- Maintenance (Experimental): Participants who usually meet or exceed recommended levels of physical activity who will be asked to maintain usual level of activity during stimulation.
  Interventions: Behavioral: Sufficient physical activity
- Usually Insufficiently Inactive- Increase (Experimental): Participants who are usually inactive who will be asked to try to increase activity to the recommended level during stimulation.
  Interventions: Behavioral: Sufficient physical activity
- Usually Insufficiently Inactive- Maintenance (Active Comparator): Participants who are usually inactive who will be asked to maintain inactivity during stimulation.
  Interventions: Behavioral: Insufficient physical activity

INTERVENTIONS:
Behavioral: Sufficient physical activity — Physical activity at the recommended levels by the US Health and Human Services Department: 75 minutes a week of vigorous activity or 150 minutes a week of moderate activity.
  Arms: Usually Active- Maintenance; Usually Insufficiently Inactive- Increase
Behavioral: Insufficient physical activity — Physical activity less than the recommended levels by the US Health and Human Services Department: 75 minutes a week of vigorous activity or 150 minutes a week of moderate activity.
  Arms: Usually Active- Decrease; Usually Insufficiently Inactive- Maintenance

SUMMARY:
Randomized control trial to determine if performing the US Health and Human Services recommended amount of weekly physical activity during ovarian stimulation will differentially affect mental health or clinical outcomes of individuals who are usually active, insufficiently active, or inactive in their everyday lives. The goal overall is to assess for safety and value of physical activity during fertility treatment.

DETAILED DESCRIPTION:
Consenting participants will be separated into groups based on current average level of physical activity: Active women (complete >75 minutes of vigorous exercise or >150 minutes of moderate exercise per week) and Insufficiently active women (<75 minutes of vigorous exercise or <150 minutes of moderate exercise per week).

Between time of study enrollment and first ultrasound at start of ovarian stimulation cycle, the participants will be sent a link to questionnaires to assess general mental health parameters and physical fitness. They will be asked to complete the questionnaire prior to first ultrasound visit. At time of first ultrasound, participants who have completed the pre-stimulation survey will be randomized into one of two arms depending on their group: the active group will be randomized to (A) maintenance or (B) decreased activity arm, and the insufficiently active group will be randomized to (C) increased or (D) maintenance activity arm.

Also at first ultrasound, participants will be given a wearable heart rate monitor in order to track heart rate during the time from ovarian stimulation to first pregnancy test in order to monitor compliance to randomized activity level of each participant. The data from the monitors will be collected through a central university provided, password protected laptop utilizing an app platform. Furthermore, all participants will be asked to complete a daily mood, stress, discomfort questionnaire throughout stimulation. Participants will be expected to continue recommended physical activity level and questionnaires until day of egg retrieval. Wearable monitors will continue to be worn until time of first pregnancy test. Within the two weeks after completion of egg retrieval, participants will be sent a follow-up questionnaire to assess overall treatment stress and satisfaction with ovarian stimulation cycle. Those who completed in vitro fertilization and fresh embryo transfer will be sent a second follow-up questionnaire about 1-2 weeks after pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* First ovarian stimulation cycle for egg freezing or for in vitro fertilization
* English speaking/reading
* Patient at the Center for Reproductive Health, University of California San Francisco

Exclusion Criteria:

* Serious health conditions that limit amount of physical activity
* BMI>40

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Stress During Treatment based on daily end of day stress item | 14 days
  As validated in prior studies (Schliep et al. 2015) examining stress and infertility, we will ask participants, "how did your stress levels today compare to your usual level of stress?" Participants will respond on a 3-point scale with the following options: 1 (not stressful), 2 (a little stressful), 3 (very stressful). We plan to compare average daily stress as well as stress trend over the 14-days of stimulation.
Anxiety/Depression During Treatment based on Patient-Reported Outcomes Measurement Information System Short Form (PROMIS-SF) Depression 4a and Anxiety 4a | 14 days
  Measured with daily PROMIS-SF Depression 4a and Anxiety 4a questions for the approximately two weeks of ovarian stimulation. The PROMIS-SF Anxiety 4a item bank assesses self-reported fear, anxious misery, hyperarousal, and arousal-related somatic symptoms (e.g., dizziness). The PROMIS-SF Depression 4a item bank assesses self-reported negative mood (e.g., sadness), views of self (e.g., worthlessness), social cognition (e.g., loneliness), and decreased positive affect and engagement. Items are all answered on a 5-point scale from 1=Never to 5=Always. Scores can range from 0 meaning no anxiety/depression to 40 meaning high anxiety/depression.
Change in Stress during treatment based upon Perceived Stress Scale (PSS)-14 | 4 weeks
  Change in mean PSS-14 score from pre-treatment to post-treatment. PSS-14 includes 14 items, 7 negatively states items and 7 positively stated items. Each item is rated on a 5-point scale (0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often). The positively stated items re reverse coded, so all items are summed to create a total score. Scores can range from 0 meaning no stress to 56 meaning severely stressed.

SECONDARY OUTCOMES:
Number of mature oocytes retrieved | 4 weeks
  Number of mature oocytes collected during oocyte retrieval after ovarian stimulation
Fertilization Rate | 4 weeks
  Number of fertilized oocytes out of the total number that were mature
Blastulation Rate | 4 weeks
  Number of blastocysts that developed out of the total number of day three embryo
Clinical Pregnancy Rate | 6 weeks
  Number of ultrasound confirmed intrauterine pregnancies out of the total ovarian stimulation cycles for in vitro fertilization
Cancellation Rate | 2 weeks
  The number of ovarian stimulation cycles that were cancelled out of all the ovarian stimulation cycles started
Ovarian Torsion | 6 weeks
  Number of ovarian torsion cases that occurred out of the total ovarian stimulation cycles
Live Birth Rate | 10 months
  Number of Live Birth out of the total ovarian stimulation cycles for in vitro fertilization
Treatment continuation rate | 4 months
  Number of women who continue treatment after first cycle if not pregnant after the first cycle

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No